CLINICAL TRIAL: NCT01447433
Title: A Randomized, Open-label, Parallel Groups-controlled Clinical Trial to Evaluate the Effect of Calcium Plus Vitamin D Supplementation on Weight Management in Overweight and Obese Very-low Calcium Consumers
Brief Title: Effect of Calcium + Vitamin D Supplementation on Weight Management in Very-low Calcium Consumers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Donglian Cai, Professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201011Z-02
Record Dates: First submitted 2011-10-04; First posted 2011-10-06 (Estimated); Results first posted 2012-03-06 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Obesity; Overweight
Keywords: Calcium Carbonate; Vitamin D; Body weight; Body fat; Metabolic parameters; Energy restriction; Very-low calcium consumers; Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight; Body Weight | interventions — Calcium Carbonate; Fumigant 93

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Calcium+D (Experimental): Calcium supplements provide 600mg of calcium and 125IU vitamin D per day. A balanced diet contains 500kcal of caloric deficit based on daily energy expenditure.
  Interventions: Drug: Calcium Carbonate; Behavioral: Energy restriction
- Control (Placebo Comparator): A balanced diet contains 500kcal of caloric deficit based on daily energy expenditure.
  Interventions: Behavioral: Energy restriction

INTERVENTIONS:
Drug: Calcium Carbonate — tablet, 600mg elemental calcium and 125IU vitamin D, once daily, for 12 weeks
  Other Names: Caltrate® 600 + D; Code:1007300
  Arms: Calcium+D
Behavioral: Energy restriction — A balanced diet contains 500kcal of caloric deficit based on daily energy expenditure.

SUMMARY:
The purpose of the study is to determine whether calcium plus vitamin D supplementation is conducive to weight and fat loss during energy restriction in very-low calcium consumers.

DETAILED DESCRIPTION:
Due to the contradicting findings in the hypothesis of calcium supplementation on weight and fat loss, which might be explained by the difference in initial calcium intake, the present study is aimed to evaluate the effect of calcium plus vitamin D supplementation on accelerating weight and fat loss in overweight or obese subjects with very-low calcium consumption(<600mg/day).

The hypotheses to be tested are:

Calcium plus vitamin D supplementation is conducive to body weight and fat loss in overweight or obese young adults during energy restriction 12 weeks after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 to 25 years of age, generally healthy
* Habitual calcium intake below 600mg/d
* Overweight or obese (BMI between 24 and 35kg/m2, refer to the Chinese standard)
* Stable body weight (body weight change less than 1kg two months before screening)
* Less than 3 times of 20min of physical exercise per week
* Signed written informed consent

Exclusion Criteria:

* Coronary heart disease, hypertension, diabetes; hepatic insufficiency or renal insufficiency, hyper- or hypothyroidism, mal-absorption, cholesterol concentrations requiring pharmaceutical treatment
* Pregnant or lactating woman
* Use of calcium supplements, oral antidiabetic agents, antihyperlipidemics or any other medications affecting metabolism 30 days before randomization
* Participating in another weight loss programs (i.e. taking oral pharmacotherapeutic agents and/or herbal preparations intended for the management of obesity; excessive physical activity; be on a diet)
* On special diets (i.e. vegetarian)
* Presently taking or have recently taken a prescription drug such as fluoroquinolone antibiotics, tetracycline, or levothyroxine (thyroid medication)
* Participating in another clinical trial 6 months before randomization
* Unlikely to be compliant (i.e. alcohol, drug abuse)
* Refusal or inability to give informed consent to participate in the study

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2011-04; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donglian Cai, Master, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, China

REFERENCES:
- [Derived] Zhu W, Cai D, Wang Y, Lin N, Hu Q, Qi Y, Ma S, Amarasekara S. Calcium plus vitamin D3 supplementation facilitated fat loss in overweight and obese college students with very-low calcium consumption: a randomized controlled trial. Nutr J. 2013 Jan 8;12:8. doi: 10.1186/1475-2891-12-8. PMID 23297844

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant were recruited through informational flyers and advertisements posted on campus of colleges and vocational schools in Pudong and Yangpu Districts in Shanghai, China. From April 20th to September 20th, 2011, a total of 129 out of 187 volunteers who answered our recruitment advertisements were invited for a pre-screening interview.
Pre-assignment Details: The pre-screening FFQ excluded 34 volunteers for habitual calcium intake>600mg/day. During screening, 16 were excluded for BMI<24kg/m2, 3 reported for using calcium supplements, 14 were on a diet, 2 refused to take calcium supplements, 1 refused to being taken blood samples, and 6 failed to sign the informed consents for personal reasons.
Period: Overall Study
Arm/Group | Calcium+D | Control
Started | 26 | 27
Completed | 22 | 21
Not Completed | 4 | 6
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Calcium+D | Control | Total
Number analyzed (Participants) | 26 | 27 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 27 | 53
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 20.3 (1.4) | 20.4 (0.8) | 20.3 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 46
  Male | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  China | 26 | 27 | 53

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight
Description: Weight was obtained in light clothing to the nearest 0.1kg using a digital scale 8:00am and 10:00am after an overnight fast between.
Time Frame: Baseline and 12 weeks
Population: Males were excluded from final analysis for statistical reasons.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Calcium+D | Control
Number analyzed (Participants) | 21 | 19
kg | -3.9 (1.7) | -3.5 (1.8)
Statistical Analysis 1: Comparison: Calcium+D vs Control; Test type: Superiority or Other; p = 0.441, t-test, 2 sided; Mean Difference (Net) = 0.439, 95% CI 2-sided [-0.70 to 1.58], Standard Error of Mean 0.56

2. Secondary Outcome: Change in Body Fat Mass，Body Lean Mass and Visceral Fat Mass
Description: BIA (bioelectric impedance analysis, ZEUS9.9, JAWON) was used to determine body fat mass, body lean mass, and visceral fat mass.
Time Frame: Baseline and 12 weeks
Population: Males were excluded from final analysis for statistical reasons.
Measure: Mean (Standard Error); unit: kg
Arm/Group | Calcium+D | Control
Number analyzed (Participants) | 21 | 19
kg
  Body Fat Mass | -2.8 (1.3) | -1.9 (1.3)
  Body Lean Mass | -0.9 (0.8) | -1.4 (0.9)
  Visceral Fat Mass | -0.47 (0.21) | -0.29 (0.21)
Statistical Analysis 1: Comparison: Calcium+D vs Control; Body Fat Mass; Test type: Superiority or Other; p = 0.038, t-test, 2 sided; Mean Difference (Net) = 0.88, 95% CI 2-sided [0.05 to 1.70], Standard Error of Mean 0.41
Statistical Analysis 2: Comparison: Calcium+D vs Control; Body Lean Mass; Test type: Superiority or Other; p = 0.082, t-test, 2 sided; Median Difference (Net) = -0.50, 95% CI 2-sided [-1.06 to 0.07], Standard Error of Mean 0.28
Statistical Analysis 3: Comparison: Calcium+D vs Control; Visceral Fat Mass; Test type: Superiority or Other; p = 0.018, t-test, 2 sided; Median Difference (Net) = 0.18, 95% CI 2-sided [0.03 to 0.32], Standard Error of Mean 0.07

3. Secondary Outcome: Change in Fat Percentage
Description: BIA (bioelectric impedance analysis, ZEUS9.9, JAWON) was used to determine fat percentage.
Time Frame: Baseline and 12 weeks
Population: Males were excluded from final analysis for statistical reasons.
Measure: Mean (Standard Deviation); unit: Percentage of body weight
Arm/Group | Calcium+D | Control
Number analyzed (Participants) | 21 | 19
Percentage of body weight | -2.6 (1.6) | -1.5 (1.5)
Statistical Analysis 1: Comparison: Calcium+D vs Control; Test type: Superiority or Other; p = 0.031, t-test, 2 sided; Median Difference (Net) = 1.10, 95% CI 2-sided [0.10 to 2.09], Standard Error of Mean 0.49

4. Secondary Outcome: Change in Visceral Fat Area
Description: BIA (bioelectric impedance analysis, ZEUS9.9, JAWON) was used to determine visceral fat area.
Time Frame: Baseline and 12 weeks
Population: Males were excluded from final analysis for statistical reasons.
Measure: Median (Standard Deviation); unit: cm^2
Arm/Group | Calcium+D | Control
Number analyzed (Participants) | 18 | 18
cm^2 | -12.5 (6.2) | -6.8 (7.2)
Statistical Analysis 1: Comparison: Calcium+D vs Control; Test type: Superiority or Other; p = 0.016, t-test, 2 sided; Median Difference (Net) = 5.72, 95% CI 2-sided [1.15 to 10.29], Standard Error of Mean 2.25

5. Secondary Outcome: Change in Waist, Abdominal and Hip Circumference
Description: Waist, abdominal and hip circumference was measured using a plastic tape to the nearest 0.1 cm
Time Frame: Baseline and 12 weeks
Population: Males were excluded from final analysis for statistical reasons.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Calcium+D | Control
Number analyzed (Participants) | 21 | 19
cm
  Waist Circumference | -6.2 (5.7) | -5.1 (5.0)
  Abdominal Circumference | -4.6 (4.4) | -5.8 (8.3)
  Hip Circumference | -4.2 (2.9) | -3.2 (2.5)
Statistical Analysis 1: Comparison: Calcium+D vs Control; Waist Circumference; Test type: Superiority or Other; p = 0.508, t-test, 2 sided; Median Difference (Net) = 1.14, 95% CI 2-sided [-2.31 to 4.58], Standard Error of Mean 1.70
Statistical Analysis 2: Comparison: Calcium+D vs Control; Abdominal Circumference; Test type: Superiority or Other; p = 0.560, t-test, 2 sided; Mean Difference (Net) = -1.22, 95% CI 2-sided [-5.42 to 2.98], Standard Error of Mean 2.07
Statistical Analysis 3: Comparison: Calcium+D vs Control; Hip Circumference; Test type: Superiority or Other; p = 0.255, t-test, 2 sided; Median Difference (Net) = 0.98, 95% CI 2-sided [-0.74 to 2.70], Standard Error of Mean 0.85

6. Secondary Outcome: Change in Blood Pressure
Description: Systolic and diastolic blood pressures were measured in the left arm at heart level of subjects seated for a minimum of 5 minutes using mercurial sphygmomanometer.
Time Frame: Baseline and 12 weeks
Population: Males were excluded from final analysis for statistical reasons.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Calcium+D | Control
Number analyzed (Participants) | 18 | 18
mm Hg
  Systolic Blood Pressure | -8.3 (13.2) | -12.1 (13.7)
  Diastolic Blood Pressure | -6.0 (9.8) | -5.0 (9.3)
Statistical Analysis 1: Comparison: Calcium+D vs Control; Systolic Blood Pressure; Test type: Superiority or Other; p = 0.404, t-test, 2 sided; Median Difference (Net) = -3.8, 95% CI 2-sided [-12.9 to 5.3], Standard Error of Mean 4.5
Statistical Analysis 2: Comparison: Calcium+D vs Control; Diastolic Blood Pressure; Test type: Superiority or Other; p = 0.768, t-test, 2 sided; Mean Difference (Net) = 0.94, 95% CI 2-sided [-5.52 to 7.41], Standard Error of Mean 3.18

7. Secondary Outcome: Change in Lipid-lipoprotein Profile
Time Frame: Baseline and 12 weeks
Population: Males were excluded from final analysis for statistical reasons.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Calcium+D | Control
Number analyzed (Participants) | 21 | 19
mmol/L
  TC | -0.11 (0.43) | -0.19 (0.45)
  TG | 0.02 (0.42) | 0.10 (0.55)
  HDL | 0.12 (0.53) | -0.14 (0.48)
  LDL | 0.14 (0.51) | 0.12 (0.40)
Statistical Analysis 1: Comparison: Calcium+D vs Control; TC; Test type: Superiority or Other; p = 0.565, t-test, 2 sided; Median Difference (Net) = -0.08, 95% CI 2-sided [-0.36 to 0.20], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: Calcium+D vs Control; TG; Test type: Superiority or Other; p = 0.636, t-test, 2 sided; Median Difference (Net) = 0.07, 95% CI 2-sided [-0.24 to 0.39], Standard Error of Mean 0.15
Statistical Analysis 3: Comparison: Calcium+D vs Control; HDL; Test type: Superiority or Other; p = 0.112, t-test, 2 sided; Median Difference (Net) = -0.26, 95% CI 2-sided [-0.58 to 0.06], Standard Error of Mean 0.16
Statistical Analysis 4: Comparison: Calcium+D vs Control; LDL; Test type: Superiority or Other; p = 0.647, t-test, 2 sided; Median Difference (Net) = -0.02, 95% CI 2-sided [-0.11 to 0.05], Standard Error of Mean 0.15

8. Secondary Outcome: Change in Fasting Plasma Glucose
Time Frame: Baseline and 12 weeks
Population: Males were excluded from final analysis for statistical reasons.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Calcium+D | Control
Number analyzed (Participants) | 21 | 19
mmol/L | 0.25 (0.33) | 0.37 (0.37)
Statistical Analysis 1: Comparison: Calcium+D vs Control; Test type: Superiority or Other; p = 0.260, t-test, 2 sided; Median Difference (Net) = 0.13, 95% CI 2-sided [-0.10 to 0.35], Standard Error of Mean 0.11

9. Secondary Outcome: Change in Fasting Plasma Insulin
Time Frame: Baseline and 12 weeks
Population: Males were excluded from final analysis for statistical reasons.
Measure: Mean (Standard Deviation); unit: mIU/L
Arm/Group | Calcium+D | Control
Number analyzed (Participants) | 21 | 19
mIU/L | -1.18 (5.02) | -0.31 (5.16)
Statistical Analysis 1: Comparison: Calcium+D vs Control; Test type: Superiority or Other; p = 0.598, t-test, 2 sided; Median Difference (Net) = 0.87, 95% CI 2-sided [-2.44 to 4.17], Standard Error of Mean 1.63

10. Secondary Outcome: Change in Energy Intakes
Time Frame: Baseline and 12 weeks
Population: Males were excluded from final analysis for statistical reasons.
Measure: Mean (Standard Deviation); unit: kcal/d
Arm/Group | Calcium+D | Control
Number analyzed (Participants) | 21 | 19
kcal/d | -400.4 (252.0) | -301.9 (310.1)
Statistical Analysis 1: Comparison: Calcium+D vs Control; Test type: Superiority or Other; p = 0.275, t-test, 2 sided; Mean Difference (Net) = 98.5, 95% CI 2-sided [-81.6 to 278.7], Standard Error of Mean 89.0

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Adverse event was assessed by questionnaires during biweekly interviews with dietitians throughout the program.
Arm/Group | Calcium+D | Control
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/27
Other Adverse Events (participants affected / at risk) | 0/26 | 0/27

LIMITATIONS AND CAVEATS:
The study sample was mostly women.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes